CLINICAL TRIAL: NCT04983381
Title: The Effect of Patient Information Training on Anxiety of Gynecologic Examination
Brief Title: Pelvic Examination Fear and Education
Acronym: [pelvicfear]
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Alime Buyuk, Principal Investigator, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2012-KAEK-20-166
Record Dates: First submitted 2021-07-12; First posted 2021-07-30 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Pelvic Pain; Pelvic Floor; Relaxation
MeSH Terms: conditions — Pelvic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education Group (Experimental): Participants were grouped as; those who were given information about vaginal examination in the training group (n=40) and those who were not given information about vaginal examination in the control group (n=40).
  Interventions: Other: Multimedia education video
- Control Group (No Intervention): Women were not given information about vaginal examination in the control group

INTERVENTIONS:
Other: Multimedia education video — The multimedia education video was a 30 minutes information-based patient education program and contained information about pelvic anatomy and how to practice vaginal examination. The same gynecologist (M.S.) (male) who 15 years of experience explained details of vaginal examination, who told about vaginal examination in this video to the study participants, also did the gynecologic examination. The gynecologic examination which contained pelvic ultrasound scan and vaginal examination lasted approximately 20 minutes practice.
  Arms: Education Group

SUMMARY:
Objectives: Gynecologic examination has been a concern for women. The aim of this study is to evaluate the effect of multimedia education on the fear of gynecologic examination.

Material and Methods: This randomized controlled study will conducted with 80 voluntary patients. Participants will grouped as training group and control group. The multimedia-based information about vaginal examination is a video based patient education program. The anxiety levels/ scores of the patients will be assessed using the State-Trait Anxiety Inventory (STAI-S [state], STAI-T [trait]) and the Visual Analog Scale (VAS). The entire evaluation will be repeated before and after the examination.

DETAILED DESCRIPTION:
The pelvic examination has been a worrisome examination for women since the initial years of gynecology science until today. Intense anxieties experienced by the patients during this examination include primarily, shame and fear of pain or pathology. Reasons such as lack of information about the gynecologic examination, previously established myths by the patient, the speculum being cold, the doctor's attitude, and the position of the examination are also among the reasons why the woman during the examination experienced anxiety. The form of gynecologic examination has varied to a large extent to this day and the examination has begun to be performed in the lithotomy position upon the invention of gynecologic examination tables. It is important that the gynecologist informs patients about the vaginal examination to be performed in this position or healthcare professionals provide short training to them. Information training typically involves the explanation of the vaginal examination and of the pelvic anatomy. The training is aimed to provide relaxation and render the examination more comfortable by explaining pelvic anatomy and pelvic floor muscles. It has been observed that these training which is provided before the interview form pelvic floor relaxation and cause less pain in the patient during the vaginal examination. Patients receiving proper and adequate training are able to understand their own complaints better and manage their disease/examination better. Patient training reduces anxiety and helps to create a more comfortable examination environment.

Previous studies have discussed patient anxieties experienced during interventions such as radiological imaging, endoscopy, colonoscopy, bronchoscopy, and invasive cardiac interventions. Short informative videos that do not cause any cost loss or harm, increase the tolerance with these applications and reduce patient anxiety. Additionally, many studies have emphasized that doctors have no time to provide information training for the vaginal examination while conducting their intense practices. Information that cannot be provided before the gynecologic examination due to limited time causes pelvic pain in women due to the anxiety experienced during the examination. The concept of chronic pelvic pain is defined as a non-cyclical pain that lasts longer than six months and develops in the pelvis and the area below the umbilicus and between the gluteal lines. Pelvic pain is observed depending on the excessive activity of pelvic floor muscles during the examination in patients who have a fear of the gynecologic examination.

The aim of this study is to evaluate the effects of multimedia education provided before the gynecologic examination on the patient's pelvic pain, anxiety, and fear.

ELIGIBILITY:
Inclusion Criteria:

* Must not have any known cerebrovascular disease,
* Must not being morbidly obese
* Must not have any heart diseases that would pose an obstacle to the study,
* Must not have any cognitive disorder that would pose an obstacle to communication,
* Must not have any stroke and the associated influence,
* Must agree to participate in the study

Exclusion Criteria:

-Reject to participate to the study

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2019-05-21 (Actual); Study Completion 2020-05-21 (Actual)

PRIMARY OUTCOMES:
Pelvic Examination of Anxiety | 6 months
  Fear about pelvic exam will be measured with Visual Analog Scale (VAS) 0 shows no fear 10 shows the most fear

CONTACTS AND LOCATIONS:
Locations (1):
- Alime Buyuk, Konyaalti, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No